CLINICAL TRIAL: NCT02429648
Title: Timing of DCC in Patients Undergoing Pulmonary Vein Isolation Ablation (PVI) of Persistent/Permanent Atrial Fibrillation
Brief Title: Timing of Direct Current Cardioversion (DCC) in Patients Undergoing Ablation of Persistent/Permanent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Walid Saliba, Walid Saliba, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09-308
Record Dates: First submitted 2010-02-01; First posted 2015-04-29 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
Keywords: AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI performed in Normal Sinus Rhythm (Active Comparator): DCC first then PVI
  Interventions: Procedure: DCC first then PVI
- PVI performed in Atrial Fibrillation (Active Comparator): PVI then DCC after if patient remains in Atrial Fibrillation
  Interventions: Procedure: PVI then DCC after

INTERVENTIONS:
Procedure: DCC first then PVI — DCC performed prior to PVI
  Arms: PVI performed in Normal Sinus Rhythm
Procedure: PVI then DCC after — DCC performed after PVI, if patient remains in Atrial Fibrillation
  Arms: PVI performed in Atrial Fibrillation

SUMMARY:
The purpose of this study is to compare which strategy is superior in patients with persistent/permanent atrial fibrillation (AF) undergoing ablation, direct current cardioversion (DCC) prior to empirical pulmonary vein isolation (PVI) ; or pulmonary vein isolation (PVI)ablation in atrial fibrillation then Direct current cardioversion (DCC) if the patient remains in atrial fibrillation.

DETAILED DESCRIPTION:
Ablation of persistent/permanent Atrial Fibrillation (AF) remains a challenge. There are several strategies to improve the outcomes of persistent/permanent AF ablation. At the Cleveland Clinic one of the commonly used strategies is Direct Current Cardioversion (DCC). Depending on physician preference, patients may be ablated in atrial fibrillation then Direct current cardioverted; or Direct current cardioverted and ablated in sinus rhythm. Neither approach has been shown to be superior. As both approaches are currently being performed based on physician preference, the investigators propose to study and compare both approaches in a randomized fashion for evidence based practice.

The purpose of this study is to compare which standard of care strategy is superior in patients with persistent/permanent Atrial Fibrillation undergoing ablation, direct current cardioversion prior to empirical pulmonary vein isolation; or ablation in atrial fibrillation then direct current cardioversion if the patient remains in atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Persistent or long standing persistent AF resistant to anti-arrhythmic medication. Must have been present for more than 2 months
* Therapeutic anticoagulation for at least three weeks prior to initiation of therapy, or TEE performed prior to the procedure
* Age >= 18 years old. (Females must be either post-menopausal >12 months, practicing a protocol-acceptable method of birth control
* Scheduled for Pulmonary Vein Isolation
* Amiodarone will be stopped at least 3 months prior to procedure

Exclusion Criteria:

* Reversible causes of AF such as pericarditis, hyperthyroidism
* Presently with Valvular Heart disease requiring surgical intervention
* Presently with coronary artery disease requiring surgical intervention
* Early Post-operative AF (within three months of surgery)
* Previous MAZE or left atrial instrumentation
* Life expectancy <= 2 years
* Social factors that would preclude follow up or make compliance difficult.
* Contraindication to the use of anti-arrhythmic medications and/or coumadin and heparin
* Enrollment in another investigational drug or device study
* Patients with severe pulmonary disease
* Documented intra-atrial thrombus, tumor, or another abnormality which precludes catheter introduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Duration of procedure | day of procedure

SECONDARY OUTCOMES:
Composite of duration of fluoroscopy, and radiation exposure doses | day of procedure
Composite of AT/AF burden and total frequency measured by event monitor, holter and/or EKG | 12 months
frequency of symptomatic atrial arrhythmias measured by event monitor, holter, and/or EKG | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Walid Saliba, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bassiouny M, Saliba W, Hussein A, Rickard J, Diab M, Aman W, Dresing T, Callahan T 4th, Bhargava M, Martin DO, Shao M, Baranowski B, Tarakji K, Tchou PJ, Hakim A, Kanj M, Lindsay B, Wazni O. Randomized Study of Persistent Atrial Fibrillation Ablation: Ablate in Sinus Rhythm Versus Ablate Complex-Fractionated Atrial Electrograms in Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2016 Feb;9(2):e003596. doi: 10.1161/CIRCEP.115.003596. PMID 26857909